CLINICAL TRIAL: NCT03296280
Title: Evaluation of Implementation of a National Point-of-Care Ultrasound Training Program
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PEX 16-003; I50HX002263-01A1 (NIH)
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Other Acute Illnesses Presenting to the Hospital; Heart Failure; Pneumonia; Deep Venous Thrombosis; Cellulitis; Abdominal Aortic Aneurysm; Acute Cholecystitis; Peritoneal Free Fluid; Hydronephrosis; Pleural Effusion; Urinary Retention
Keywords: ultrasound; ultrasonography; point of care; Doppler ultrasound; ultrasound imaging; diagnostic ultrasound
MeSH Terms: conditions — Heart Failure; Pneumonia; Venous Thrombosis; Cellulitis; Aortic Aneurysm, Abdominal; Cholecystitis, Acute; Hydronephrosis; Pleural Effusion; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Early Intervention: This cohort of 10 facilities will undergo early training by participating in the first 6 POCUS course sessions during FY17
- Late Intervention: This cohort of 10 facilities will undergo late training by participating in the last 6 POCUS courses during FY17.

SUMMARY:
This VA QUERI Partnered Evaluation Initiative will evaluate the impact of an immersive Point-of-care Ultrasound (POCUS) Training Course on provider skill acquisition and retention; the frequency of POCUS use by trained providers; and the barriers/facilitators to POCUS in the VHA. Data sources include pre- and post-course assessment tools, medical coding data, and course evaluations. Providers that participate in the POCUS Training Course will be compared to control providers from wait-listed facilities. Additionally, participating facilities vs. wait-listed facilities for the POCUS Training Course will be compared. Findings from this project will guide ongoing efforts of the investigators' operating partners, VA Specialty Care Centers of Innovation (SCCI) and the VA Simulation Learning and Research Network (SimLEARN), to develop a national POCUS training program and facilitate implementation of POCUS use system-wide in the VA healthcare system.

DETAILED DESCRIPTION:
Background: Point-of-care ultrasonography (POCUS) has been shown to reduce procedure-related complications from invasive bedside procedures, reduce time to diagnosis, and reduce ancillary testing, which ultimately reduces patient radiation exposure and healthcare costs. Despite its potential advantages, POCUS has not been universally adopted in healthcare due to limited numbers of providers trained in use of POCUS. The VA's Simulation Learning, Education and Research Network (SimLEARN) and Specialty Care Centers of Innovation (SCCI) have launched a collaborative initiative to develop a national POCUS training program. The goal of this collaborative training program is to teach VA providers basic diagnostic and procedural applications of POCUS. The proposed project will evaluate the effectiveness of an immersive POCUS training course developed by SimLEARN on provider skill acquisition and retention, frequency of use, and identify barriers/facilitators to POCUS use at participating VHA facilities.

Methods: Approximately 120 participants from a convenience sample of 20 diverse VA facilities will participate in a 2.5-day immersive POCUS training course at the SimLEARN National Simulation Center in Orlando during fiscal year 2017. The investigators' evaluation plan will collect data from facility Chiefs of Staff, providers from facilities participating in POCUS training, and providers from wait-listed facilities at different time points using different assessment tools: VA Facility POCUS Survey, Provider POCUS Survey, Brief Provider POCUS Survey, Pre-/Post-course Knowledge and Skills Test, and Coding Data.

Objective 1: Evaluate provider skill acquisition and retention, and frequency of POCUS use after participation in the POCUS Training Course. Pre- and post-course testing will be used to assess acquisition of knowledge and technical skills to perform POCUS exams. Post-course testing for knowledge and skill retention, and frequency of use, will be performed 6-9 months after the training course.

Objective 2: Determine the effect of the POCUS Training Course and implementation facilitation on facility-level frequency of POCUS use. Facilities with providers that infrequently use POCUS will be eligible to participate in the POCUS Training Course. However, not all facilities will be able to be accommodated in the 1st year of the training program, requiring a facility waiting list. Facilities with providers participating in the POCUS Training Course will be compared to wait-listed facilities with regard to frequency of POCUS use. Using the Brief Provider POCUS Survey, frequency of POCUS use by providers in both participating and waitlisted facilities will be compared. Additionally, coding data will be reviewed to assess frequency of procedures performed with and without imaging guidance and procedural complication rates comparing the two groups of facilities.

Objective 3: Determine provider and facility-level barriers and facilitators to POCUS use. Provider and facility-level barriers will be assessed using 3 tools: Provider POCUS Survey (trained providers), Brief Provider POCUS Survey (wait-listed and participating facilities), and Facility POCUS Survey (all facilities). Differences in barriers reported and their relationship to frequency of POCUS use will be compared.

Objective 4: Development of POCUS Champions course to facilitate local implementation by addressing facility-level barriers. The POCUS Champions course will address several facility-level barriers to implementation that have been identified by the PEI: lack of image archiving, limited access to ultrasound machines, undefined credentialing/privileging processes, need for a quality assurance process, and lack of trained providers. The POCUS Champions course will include an annual 3-day boot camp, bi-monthly conference calls, and ongoing mentorship. The goal of the 3-day boot camp will be for Champions to prepare a local implementation plan that can be presented to their facility's leadership. During the bimonthly conference calls, a brief didactic on a focused topic will be presented followed by an update on local progress from each site. The initial goal of the POCUS Champions course is to facilitate implementation of POCUS use in VA facilities, starting with 4-6 facilities that can serve as models for other facilities. The research to date has identified these elements as core components of a successful POCUS program. The POCUS Champions course will support progress on intermediate milestones towards ensuring these core components are in place, to facilitate adoption, reach, and sustainment. This provides a roadmap to sustainable POCUS use.

Deliverables: The primary deliverable will be report that will summarize the effect of training on provider skill acquisition and retention, frequency of use of POCUS, and barriers and facilitators to POCUS implementation. This project will guide SimLEARN's and SCCI's efforts to develop a National POCUS Training Program and implement POCUS use nationally in the VA healthcare system. Additionally, this report may serve as a roadmap for the VHA for implementation of similar simulation-based educational innovations.

ELIGIBILITY:
Inclusion Criteria:

Selection of VA facilities invited to participate in the national POCUS training course was based on data from a national needs assessment conducted by the VA's Health Analysis and Information Group. VA facilities that meet all of the following inclusion criteria are eligible to send physicians to participate in the POCUS training course:

1. Chief of staff desires POCUS training for his/her facility
2. >=2 Service Chiefs from emergency medicine, critical care medicine, or hospital medicine desire training for his/her physicians, AND
3. >=1 portable ultrasound machine(s) available to physicians within these services

Exclusion Criteria:

1. Chief of staff does not desire POCUS training for his/her facility
2. <2 Service Chiefs from emergency medicine, critical care medicine, or hospital medicine desire training for his/her physicians, OR
3. No portable ultrasound machine(s) available to physicians within these services

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: VA physicians
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilam Jayant Soni, MD MSc, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iqbal A, Ahmad M, Murray KJ, Sim J, Lund TJS, Andrade AJ, Perez-Sanchez A, Mader MJ, Haro EK, Williams JP, Nathanson R, Soni NJ. Current Use and Barriers to Point-of-Care Ultrasound in Rheumatology: A National Survey of VA Medical Centers. Rheumatol Ther. 2024 Jun;11(3):855-867. doi: 10.1007/s40744-024-00665-2. Epub 2024 Apr 6. PMID 38581600
- [Derived] Boyd JS, LoPresti CM, Core M, Schott C, Mader MJ, Lucas BP, Haro EK, Finley EP, Restrepo MI, Kessler C, Colon-Molero A, Pugh J, Soni NJ. Current use and training needs of point-of-care ultrasound in emergency departments: A national survey of VA hospitals. Am J Emerg Med. 2019 Sep;37(9):1794-1797. doi: 10.1016/j.ajem.2019.02.043. Epub 2019 Feb 28. No abstract available. PMID 30878406
- See also: VA Quality Enhancemen Research Initiative (QUERI) — https://www.queri.research.va.gov/national_partnered_evaluations/ultrasound.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 facilities were to participate in the first 6 POCUS course session during FY17. 10 facilities were to participate in the last 6 POCUS course sessions during FY17. Participants, rather than facilities, were recruited and assigned to to the early or late intervention arms.
Groups:
- Early Intervention: This cohort of 10 facilities will undergo early training by participating in the first 6 POCUS course sessions during FY17. Although facilities are being recruited the intervention is taking place at the individual level. All reporting will be at the individual level.
- Late Intervention: This cohort of 10 facilities will undergo late training by participating in the last 6 POCUS courses during FY17. Although facilities are being recruited the intervention is taking place at the individual level. All reporting will be at the individual level.
Period: Overall Study
Arm/Group | Early Intervention | Late Intervention
Started | 73 | 43
Completed | 67 | 36
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Intervention | Late Intervention | Total
Number analyzed (Participants) | 73 | 43 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row populations differs from Overall because age was self-reported through an online survey and was not answered by all participants.
  years
    number analyzed (Participants) | 70 | 39 | 109
    (all) | 45.7 (10.6) | 43.5 (7.7) | 44.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row populations differs from Overall because sex was self-reported through an online survey and was not answered by all participants.
  Participants
    number analyzed (Participants) | 70 | 39 | 109
    Female | 27 | 18 | 45
    Male | 43 | 21 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Provider Specialty [Number; unit: participants] — Population: Row populations differs from Overall because provider specialty was self-reported through an online survey and was not answered by all participants.
  participants
    Anesthesiology: number analyzed (Participants) | 70 | 39 | 109
    Anesthesiology | 6 | 7 | 13
    Critical Care: number analyzed (Participants) | 70 | 39 | 109
    Critical Care | 10 | 8 | 18
    Emergency Medicine: number analyzed (Participants) | 70 | 39 | 109
    Emergency Medicine | 13 | 9 | 22
    Endocrinology: number analyzed (Participants) | 70 | 39 | 109
    Endocrinology | 1 | 0 | 1
    General Surgery: number analyzed (Participants) | 70 | 39 | 109
    General Surgery | 0 | 3 | 3
    Internal Medicine: number analyzed (Participants) | 70 | 39 | 109
    Internal Medicine | 31 | 10 | 41
    Pulmonary: number analyzed (Participants) | 70 | 39 | 109
    Pulmonary | 8 | 2 | 10
    Other: number analyzed (Participants) | 70 | 39 | 109
    Other | 1 | 0 | 1
Facility Location [Number; unit: participants]
  Continental | 13 | 0 | 13
  Midwest | 11 | 4 | 15
  Northeast | 8 | 12 | 20
  Pacific | 11 | 11 | 22
  Southeast | 30 | 16 | 46
Years of practice since residency [Mean (Standard Deviation); unit: years] — Population: Row populations differs from Overall because years since residency was self-reported through an online survey and was not answered by all participants.
  years
    number analyzed (Participants) | 70 | 39 | 109
    (all) | 14.8 (10.4) | 11.5 (6.9) | 13.6 (9.5)
Percent of time performing direct patient care [Mean (Standard Deviation); unit: % of time performing direct pt care] — Population: Row populations differs from Overall because percent of time performing direct patient care was self-reported through an online survey and was not answered by all participants.
  % of time performing direct pt care
    number analyzed (Participants) | 70 | 39 | 109
    (all) | 57 (30) | 58 (23) | 57 (28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Point-of-care Ultrasound Use for Diagnostic and Procedural Applications at Baseline and 6-9 Months
Description: Provider self-reported data pre- and post-intervention on frequency of point-of-care ultrasound use, based on number of exams per week.
Time Frame: Baseline compared to 6-9 months later.
Population: Participants who completed a provider survey both at the start and about 6-9 months later
Measure: Mean (95% Confidence Interval); unit: Number of POCUS Exams/week
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 62 | 33
Number of POCUS Exams/week | 12.9 [4.5 to 21.3] | 4.0 [1 to 7]

2. Secondary Outcome: Change in Point-of-care Ultrasound Knowledge From Baseline to 6-9 Months
Description: Provider knowledge will be tested pre- and post-intervention (at baseline [pre-course] and 6-9 months post-course). Knowledge Exam has a minimum of 0 points and a maximum of 30 points (1 pt per question). A higher score indicates more knowledge about POCUS. A positive change in score means a better outcome post-course (net increase in knowledge) compared to baseline.
Time Frame: Baseline compared to 6-9 months later.
Population: Participants who completed a knowledge survey both at the start and about 6-9 months later were analyzed. Those who did not provide both surveys are not reported. Row populations may therefore differ from total population counts.
Measure: Mean (95% Confidence Interval); unit: change in score on POCUS Knowledge scale
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 57 | 27
change in score on POCUS Knowledge scale | 5.3 [4.4 to 6.2] | 6.5 [4.4 to 8.6]

3. Secondary Outcome: Change in Point-of-care Ultrasound Cardiac Skills From Baseline to 6-9 Months
Description: Provider hands-on cardiac skills will be tested pre- and post-intervention (at baseline [pre-course], and 6-9 months post-course). The minimum score on the POCUS Cardiac Skills scale is 0 points and the maximum is 100 points. A higher score indicates more skill. A positive change in score means a better outcome post-course (net increase in skills) compared to baseline.
Time Frame: Baseline compared to 6-9 months later.
Population: Participants who completed a skills survey both at the start and about 6-9 months later were analyzed. Those who did not provide both surveys are not reported. Row populations may therefore differ from total population counts.
Measure: Mean (95% Confidence Interval); unit: change in score on Cardiac Skills scale
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 58 | 23
change in score on Cardiac Skills scale | 41.6 [35.2 to 48.0] | 46.1 [35.6 to 56.6]

4. Secondary Outcome: Change in Point-of-care Ultrasound Lung Skills From Baseline to 6-9 Months
Description: Provider hands-on lung skills will be tested pre- and post-intervention (at baseline [pre-course], and 6-9 months post-course). The minimum score on the POCUS Lung Skills scale is 0 points and the maximum is 100 points. A higher score indicates more skill. A positive change in score means a better outcome post-course (net increase in skills) compared to baseline.
Time Frame: Baseline compared to 6-9 months later.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: change in score on Lung Skills scale
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 58 | 24
change in score on Lung Skills scale | 49.2 [43.4 to 55.0] | 60.5 [50.8 to 70.3]

5. Secondary Outcome: Change in Point-of-care Ultrasound Peripheral IV Skills From Baseline to 6-9 Months
Description: Provider hands-on peripheral IV skills will be tested pre- and post-intervention (at baseline [pre-course], and 6-9 months post-course). The minimum score on the POCUS Peripheral IV Skills scale is 0 points and the maximum is 100 points. A higher score indicates more skill. A positive change in score means a better outcome post-course (net increase in skills) compared to baseline.
Time Frame: Baseline compared to 6-9 months later.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: change in score on Peri-IV Skills scale
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 54 | 21
change in score on Peri-IV Skills scale | 31.6 [24.7 to 38.6] | 40.5 [26.1 to 54.9]

6. Secondary Outcome: Change in Point-of-care Ultrasound Abdominal Skills From Baseline to 6-9 Months
Description: Provider hands-on abdominal skills will be tested pre- and post-intervention (at baseline [pre-course], and 6-9 months post-course). The minimum score on the POCUS Abdominal Skills scale is 0 points and the maximum is 100 points. A higher score indicates more skill. A positive change in score means a better outcome post-course (net increase in skills) compared to baseline.
Time Frame: Baseline compared to 6-9 months later.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: change in score on Abdom Skills scale
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 58 | 24
change in score on Abdom Skills scale | 40.8 [34.1 to 47.5] | 54.8 [44.7 to 65.0]

7. Secondary Outcome: Change in Barrier to Point-of-care Ultrasound Use (Ability to Operate) From Baseline to 6-9 Months Post-Course
Description: Change in percentage of providers who reported not knowing how to operate POCUS 6-9 months post-course compared to pre-course. A positive percentage indicates a better outcome post-course.
Time Frame: Baseline compared to 6-9 months later.
Population: Participants who reported not knowing how to use POCUS machine in survey at the beginning of the course
Measure: Number; unit: percentage of participants
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 22 | 9
percentage of participants | 68 | 67

8. Secondary Outcome: Change in Barriers to Point-of-care Ultrasound Use (Skill Maintenance) From Baseline to 6-9 Months Post-Course
Description: Change in percentage of providers who reported experiencing difficulty with maintaining POCUS skills pre-course compared to 6-9 months post-course. A positive percentage indicates more providers are experiencing this barrier post-course, which is not unexpected as more providers acquire POCUS skills.
Time Frame: Baseline compared to 6-9 months later.
Population: Participants who reported at least one barrier 6-9 months after course
Measure: Number; unit: percentage of participants
Arm/Group | Early Intervention | Late Intervention
Number analyzed (Participants) | 30 | 19
percentage of participants | 23 | 37

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored. Not applicable.
Description: Adverse events were not monitored. Not applicable.
Arm/Group | Early Intervention | Late Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Maintaining early or late intervention groups due to schedules/space limitations.
2. Equipment not readily available and inability to receive IT approvals limited follow-up scheduling.
3. Participants with limited clinical time may skew scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03296280/Prot_SAP_000.pdf